CLINICAL TRIAL: NCT05035420
Title: A Pilot Study to Evaluate A Noninvasive Multimodal Biosensing Device for Screening and Monitoring Response to Treatment of Infectious Respiratory Diseases
Brief Title: A Noninvasive Multimodal Biosensing Device for Screening and Monitoring Response to Treatment of Infectious Respiratory Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 210028; 21-CH-0028
Record Dates: First submitted 2021-09-03; First posted 2021-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09-03

CONDITIONS: COVID-19; Upper Respiratory Infection; Lower Respiratory Infection
Keywords: point-of-care multimodal biosensing device; COVID-19 screening and monitoring
MeSH Terms: conditions — COVID-19; Respiratory Tract Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteer (Experimental): Healthy Volunteer
  Interventions: Device: Fitbit; Device: Douglas Bag; Device: Periflux 6000 EPOS; Device: BIOPAC; Device: Flowmet; Device: NIRS

INTERVENTIONS:
Device: Fitbit — Performance of the NIRS biosensor will be explored in comparison to this commercial wearable.
Device: Douglas Bag — The Douglas Bag will be used for inducing hypercapnia.
Device: Periflux 6000 EPOS — Tissue oxygen saturation measured by the Periflux 6000 will be compared with peripheral tissue saturation measured with the NIRS biosensor both at rest and during the induced hypercapnia, paced breathing and breath holding.
Device: BIOPAC — The BIOPAC system will be used to record the PPG signal, cardiovascular hemodynamics, and respiratory parameters in order to noninvasively monitor the heart rate, heart rate variability, respiratory rate, respiratory effort index, and arterial oxygen saturation.
Device: Flowmet — Flowmet will be used for a measurement of arterial blood flow within the finger or toe. Flowmet outputs a PPG waveform that will be compared with the NIRS biosensor.
Device: NIRS — a. Each subject will be monitored with the multimodal system for 10 minutes while sitting quiescent on a chair in resting position. All screening index parameters will be collected and recorded. b. Each subject will be studied for approximately 60-80 minutes while being exposed to a mild Hypercapnia (5% CO2), paced breathing and breath holding followed by a 10-minute recovery time after each task.

SUMMARY:
Background:

The COVID-19 outbreak has strained the health care system. New tools are needed for diagnostic testing and monitoring of people who have the virus. Researchers want to test a device they hope can screen, detect, and monitor symptoms linked to respiratory diseases like COVID-19.

Objective:

To evaluate and validate a device that measures breathing, body temperature, heart rate, and tissue oxygenation.

Eligibility:

Healthy adults ages 18 and older with no flu-like symptoms and no current signs of infection, cough, fever, or sneezing.

Design:

Participants will have a physical exam. Their vital signs will be taken.

Participants will sit in a chair. They will be monitored for 60 to 80 minutes while they do the following tasks:

Rest for 10 minutes. They will repeat this after each task.

Hold their breath for up to 2 minutes and then rest for 2 minutes. They will do this task 3 times.

Pace-breathe with breathing rates of 10, 20, and 30 breaths per minute. They will do this task 2 times.

Breathe air that has 5% of carbon dioxide for 5 minutes.

During these tasks, data will be collected and recorded with a pulse oximeter, thermometer, respiratory belt, and spirometer.

Participants will fill out questionnaires related to their daily activity (medication intake, exercise, smoking, and drinking).

Participation will last for 2 to 3 hours.

DETAILED DESCRIPTION:
Study Description:<TAB>

This observational pilot study will characterize the performance of a multimodal biosensor device (a portable and a wireless NIRS device, PPG and temperature sensor) in measuring human vital signs, which later will be explored as a point-of-care method for screening and treatment response monitoring of individuals with an infectious respiratory illness. The devices will measure heart, respiratory, and tissue oxygenation parameters in healthy subjects at rest and during induced hypercapnia, breath holding, and paced breathing.

Objectives:

<TAB>

Primary objective: Compare performance of two multimodal NIRS biosensor devices with commercial systems for measuring vital physiological signals including cardiac, respiratory, and tissue oxygenation in individuals at rest.

Secondary objective: Compare measured changes in cardiac, respiratory, and tissue oxygenation parameters during induced hypercapnia, breath holding, and paced breathing exercises between the biosensor and commercial systems.

Exploratory objective: Characterize arterial oxygen saturation (SpO2), peripheral oxygen saturation (StO2) and cerebral oxygen saturation (ScO2) during respiratory perturbations.

Endpoints:<TAB>

Primary endpoint: Paired differences, Lin s concordance correlation coefficient and Bland-Altman analysis for the following parameters: Biosensor tissue microvascular oxygenation level (StO2), respiratory rate (RR), respiratory effort index (REI), heart rate (HR) and heart rate variability (HRV).

Secondary endpoint: Paired differences, Lin s concordance correlation coefficient and Bland-Altman analysis for the following parameters: Biosensor tissue microvascular oxygenation level (StO2), respiratory rate (RR), respiratory effort index (REI), heart rate (HR) and heart rate variability (HRV) during induced hypercapnia, breath holding, and paced breathing exercises.

Exploratory endpoint: Arterial oxygen saturation (SpO2), peripheral oxygen saturation (StO2) and cerebral oxygen saturation (ScO2).

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Provision of signed and dated informed consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female aged 18 years or greater.
* In good general health as evidenced by medical history with no signs of cough, sneeze and upper respiratory symptoms.
* Body temperature in normal range (afebrile, temperature < 100.4 (Infinite) F) on the day of the experiment.

EXCLUSION CRITERIA:

* Any skin disease.
* Fever (Temperature greater than or equal to 100.4 degrees F).
* Any past or present cardiovascular or pulmonary diseases.
* Known adverse reaction to latex.
* Any medical condition that, in the opinion of the Principal Investigator would preclude the inclusion of a patient onto this research study.
* Unable or unwilling to give informed consent.
* Individuals with known respiratory conditions.
* Individuals who are currently taking medication that may cause methemoglobinemia such as nitrates derivatives, sulfonamides, dapsone, phenacetin, phenazopyridine, some local anesthetics such as prilocaine, topical anesthetics such as emla cream, benzocaine.
* Individuals with history of seizure.
* Smokers and those on narcotics.
* Pregnant women are excluded due to risk associated to hypercapnia risk

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Compare performance of a multimodal biosensor device with commercial systems for measuring vital physiological signals including cardiac, respiratory, and tissue oxygenation in individuals at rest. | End of study
  Compare performance of two multimodal NIRS biosensor devices with commercial systems for measuring vital physiological signals including cardiac, respiratory, and tissue oxygenation in individuals at rest.

SECONDARY OUTCOMES:
Characterize arterial oxygen saturation (SpO2), peripheral oxygen saturation (StO2) and cerebral oxygen saturation (ScO2) during respiratory perturbations. | End of study
  We would like to know if arterial oxygen saturation (SpO2), peripheral oxygen saturation (StO2) and cerebral oxygen saturation (ScO2) are also sensitive to respiratory changes. Although these parameters are all related, they may exhibit unique behavior due to autoregulatory mechanisms in the brain and differences between arterial and tissue saturation.
Compare measured changes in cardiac, respiratory, and tissue oxygenation parameters during induced hypercapnia, breath holding, and paced breathing exercises between the biosensor and commercial systems. | End of study
  Accuracy of the biosensor not only depends on comparison to baseline values but also should correlate during induced changes.

CONTACTS AND LOCATIONS:
Overall Officials: Amir H Gandjbakhche, Ph.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
We are working on deciding if we will share IPD

REFERENCES:
- [Background] Sakudo A. Near-infrared spectroscopy for medical applications: Current status and future perspectives. Clin Chim Acta. 2016 Apr 1;455:181-8. doi: 10.1016/j.cca.2016.02.009. Epub 2016 Feb 12. PMID 26877058
- [Background] Chiu WT, Lin PW, Chiou HY, Lee WS, Lee CN, Yang YY, Lee HM, Hsieh MS, Hu CJ, Ho YS, Deng WP, Hsu CY. Infrared thermography to mass-screen suspected SARS patients with fever. Asia Pac J Public Health. 2005;17(1):26-8. doi: 10.1177/101053950501700107. PMID 16044829
- [Background] Abay TY, Kyriacou PA. Reflectance Photoplethysmography as Noninvasive Monitoring of Tissue Blood Perfusion. IEEE Trans Biomed Eng. 2015 Sep;62(9):2187-95. doi: 10.1109/TBME.2015.2417863. Epub 2015 Mar 30. PMID 25838515
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2021-CH-0028.html